CLINICAL TRIAL: NCT03069235
Title: Operational Research to Promote Breastfeeding Among HIV Infected Women Attending the Prevention of Mother to Child Transmission (PMTCT) Program in Mulago Hospital, Kampala, Uganda
Brief Title: Promoting Exclusive Breastfeeding Among HIV Infected Women in a PMTCT Program
Acronym: EBF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: MU-JHU CARE (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NA_00050616
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: HIV-infection/Aids; Breast Feeding
Keywords: HIV; Breast Feeding
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Breast Feeding | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (Active Comparator): group/individual counselling.
  Interventions: Behavioral: standard of care
- Family member / peer support (Experimental): Structured family member / peer support.
  Interventions: Behavioral: Family member / peer support
- Special infant feeding counselor support (Experimental): Enhanced intervention with counselor support
  Interventions: Behavioral: Family member / peer support; Behavioral: Enhanced intervention with counselor support

INTERVENTIONS:
Behavioral: Family member / peer support — supplemental individualized counselling
  Arms: Family member / peer support; Special infant feeding counselor support
Behavioral: Enhanced intervention with counselor support — "hands on" EBF demonstrations
  Arms: Special infant feeding counselor support
Behavioral: standard of care — one on one and in-group counselling
  Arms: Standard of Care

SUMMARY:
This study evaluates strategies aimed at promoting exclusive breast feeding for 6 months followed by continued breastfeeding for the next 6 months with introduction of complementary foods among HIV infected women in a resource limited setting.

DETAILED DESCRIPTION:
This is a single center, operational research study with two components. A formative component and randomized intervention trial. The study aims are to inform, promote and evaluate strategies aimed at promoting exclusive breast feeding for 6 months followed by continued breastfeeding for the next 6 months with introduction of complementary foods among HIV infected women in a resource limited settings.

The primary objective of the qualitative formative research which includes Focus Group Discussions (FGD) and Key Informant Interviews (KII) is to explore factors affecting decisions on EBF and continued breastfeeding among HIV infected women.

The primary objective for the Intervention phase is to compare either of two intervention strategies against the standard arm using Ministry of Health (MOH) messages aimed at promoting EBF for 6 month.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive pregnant women in their late second or third trimester
* On antiretroviral therapy (ARVs) for PMTCT or meets MOH guidelines for ARV therapy
* Intention to breast feed
* Willingness to deliver at Mulago Hospital
* Living within Kampala and planning to stay within Kampala district for months after delivery
* Willingness to participate during post partum period
* Willingness to be home visited
* Willingness and ability to bring a close family member of choice to the clinic, who is ≥ 18 years, who will be able to be in touch with the at least three times a week and to give support on EBF

Exclusion Criteria:

* none

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 218 (Actual)
Dates: Start 2012-02-08 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2013-11-30 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding | six months
  proportion of women who report exclusive breastfeeding to six months

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Matovu, MA, Principal Investigator — MU-JHU CARE

IPD SHARING:
Plan to Share IPD: No